CLINICAL TRIAL: NCT06495710
Title: Load-Dependent Arterial Stiffness to Optimize Blood Pressure Management in Older Veterans (LOADED BP)
Brief Title: Arterial Stiffness and Blood Pressure
Acronym: LOADED-BP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Tennessee Valley Health Care System (U.S. Federal Agency); Birmingham, Alabama VA Medical Center (U.S. Federal Agency); The Lundquist Institute (Unknown); University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CARB-007-23F
Record Dates: First submitted 2024-05-24; First posted 2024-07-11 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Hypertension; Vascular Stiffness; Aging
Keywords: hypertension; Vascular Stiffness; Aging
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intensive BP targets (Experimental): <120 mmHg systolic)
  Interventions: Other: Blood pressure treatment algorithm
- Standard blood pressure targets (Active Comparator): <140 mmHg systolic
  Interventions: Other: Blood pressure treatment algorithm

INTERVENTIONS:
Other: Blood pressure treatment algorithm — Single or combination antihypertensive therapy as needed: 1) amlodipine (2.5-10 mg), 2) telmisartan (20-80 mg) or losartan (25-100 mg), 3) chlorthalidone (6.25-25 mg), or 4) spironolactone (12.5-50 mg). a two-drug regimen with either amlodipine + chlorthalidone or telmisartan + chlorthalidone will be initiated following randomization. If a diuretic is contraindicated, amlodipine + telmisartan will be initiated. For those over 75 years, either amlodipine or telmisartan will be initiated at baseline if SBP is <140 mmHg. In the standard treatment group (SBP goal of < 140 mmHg), participants will either be prescribed amlodipine or telmisartan/losartan as initial therapy. If >3 medications are necessary to reach the intensive goal and no first line options remain, potassium sparing diuretics or direct vasodilators will be considered.

SUMMARY:
Hypertension is a common and treatable disorder that remains the leading preventable cause of heart disease. Blood pressure treatment relies mainly on upper arm blood pressure readings and ignores blood vessel physiology and underlying individual genetic information. Older Veterans with hypertension are less likely to be treated to goal blood pressure because there are conflicting recommendations for what constitutes "optimal" in older adults. The investigators have developed a novel way to non-invasively assess the components of blood vessel stiffness that is related to blood pressure (load-dependent stiffness). This project will generate new knowledge about how different blood pressure treatment goals (intensive vs standard) impact different components of arterial stiffness and if these differences can be explained through genetic analysis. Results from this project will offer the VA an updated blueprint for personalizing blood pressure care in older adults, ultimately improving cardiovascular health.

DETAILED DESCRIPTION:
Aims and Rationale: Hypertension is ubiquitous within the VA system and is the leading cause of preventable cardiovascular disease in the United States. Over 1/3 of Veterans with hypertension are not treated to goal, and there are significant differences between professional guideline statement recommendations. A critical knowledge-practice gap exists in blood pressure (BP) management: Treatment decisions in older adults rely mainly on brachial artery BP measurements, ignoring arterial stiffness mechanisms and the underlying genetics of hypertension. The investigators need non-invasive tools to identify older adults most likely to benefit from more intensive BP targets. The investigators plan to evaluate novel physiologic mechanistic arterial stiffness measures (load-dependent stiffness and structural stiffness) and a known BP polygenic risk score (PRS) to improve hypertension care in older Veterans. Total arterial stiffness (e.g., arterial wall rigidity) has two distinct components: 1) structural stiffening due to arterial wall remodeling (e.g., elastin degradation and fibrin and collagen deposition) and 2) load-dependent stiffness, by which elevated BP increases collagen fiber loading. The investigators hope to use these tools to improve the understanding of individual differences in BP treatment responses. The investigators plan to determine if intensive vs. standard BP treatment (i.e., <120 vs. <140 mmHg) improves arterial stiffness components (load-dependent and structural) in older hypertensive Veterans with baseline systolic BP 140 mmHg) over 12 months and determine if baseline load dependent stiffness is associated with BP response regardless of treatment group. Finally, the investigators will determine if a BP PRS can be used to explain individual variability in stiffness responses. A straightforward non-invasive arterial stiffness test, like load dependent stiffness, combined with genetic markers, could improve hypertension and CVD outcomes by personalizing treatment plans in this at-risk Veteran demographic.

Methods: The investigators propose a three-site randomized controlled trial that will enroll hypertensive Veterans 60 years old (n=228). Participants will be randomized 1:1 to intensive or standard BP treatment (<120 vs <140 mmHg). The primary outcomes of load-dependent and structural arterial stiffness will be assessed at baseline and after 3, 6 and 12 months of guideline-based antihypertensive therapy. Medications will be prescribed and titrated at each visit, and serious adverse effects including hypotension, acute kidney injury and falls will be documented. This will permit the analysis of the impact of BP treatment goals of the mechanistic components of arterial stiffness in older Veterans (primary outcome) and improve the understanding of the underlying genetic factors related to the individual differences in stiffness mechanisms and their specific BP response to treatment goals.

Innovation/Significance: BP control is a major unaddressed problem in the VA Health system. Load-dependent arterial stiffness measures and a BP PRS may provide a novel way to personalize BP goals in older adults and offer new insights into complex phenotypic and genetic differences in BP response. The interaction between blood pressure and stiffness is well described for total arterial stiffness measures, but the impact of standard vs. intensive blood pressure targets on both phenotypic arterial stiffness (load-dependent vs structural stiffness) and genotypic associations with a blood pressure specific polygenic risk score (PRS) has not been studied in older adults. This non-invasive stiffness test could be used as a novel risk-stratification tool to help identify older patients who would benefit from the most aggressive BP treatment goals, ultimately decreasing CVD events in this at-risk population. This will facilitate further studies that could eventually lead to the use of these techniques in clinical settings, allowing prescribers to easily and non-invasively identify older Veterans at the highest CVD risk and more easily assign optimal blood pressure targets to each patient.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants from VA VISN 7, 9, and 12 will be eligible to participate if they are over age 60 years and have a diagnosis of hypertension or take antihypertensive medications (up to 4).
* Veterans will require documented SBP readings on 2 or more office visits that are 140 mmHg or average home blood pressure readings 135 mmHg to be eligible for the trial.
* Participants must be willing to be randomized to intensive or standard blood pressure treatment and have blood pressure medications adjusted per the study protocol.
* They must be willing to undergo tonometric evaluation of arterial stiffness, and carotid artery ultrasound.

Exclusion Criteria:

* Participants who have an indication for a specific BP lowering medication that is not included in the study protocol or a known secondary cause of hypertension will be excluded.
* Patients will be excluded if they have:

  * a standing SBP <110 mmHg
  * past history of a recent CVD event in the past 12 months (i.e., coronary artery disease event/intervention, congestive heart failure exacerbation or heart failure hospitalization, atrial fibrillation, or peripheral arterial disease intervention)
  * a class I indication for betablocker use including atrial arrhythmias
  * left-ventricular systolic function <50%, >moderate aortic stenosis
  * history of stroke
  * chronic kidney disease (eGFR<30 mL/min/m2) or proteinuria in excess of 1 gram/day or polycystic kidney disease
  * active cancer (other than untreated, non-metastatic prostate cancer and non-melanoma skin cancer)
  * hypoxemic pulmonary disease
  * active rheumatologic or connective tissue diseases (i.e., systemic lupus erythematosus, rheumatoid arthritis, etc.)
  * human immunodeficiency virus
  * illness with any infectious etiology or fever >38°C (i.e., upper respiratory illness, gastrointestinal illness, etc.)
  * hospitalization for any reason within the prior 4 weeks
* Participants will be excluded if arm circumference is too large/small to allow accurate blood pressure recordings
* The investigators will also exclude those with factors that may limit adherence to the study interventions or follow-up including active substance abuse, plans to move outside the study catchment areas within 12 months or a history of poor medication adherence or clinic no-shows

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Load-dependent arterial stiffness measured with pulse wave velocity (m/s) | 12 months
  Load dependent stiffening is measured with ultrasound and tonometry and is the stiffness component due to elevated blood pressure increasing collagen fiber loading without an intrinsic change to the artery wall. The primary outcomes of load-dependent stiffness will be assessed at baseline and after 3, 6 and 12 months of guideline-based antihypertensive therapy.
Structural arterial stiffness measured with pulse wave velocity (m/s) | 12 months
  Structural stiffening is measured with ultrasound and tonometry and is the stiffness component due to growth (eg. intima-media thickening) and remodeling (eg. elastin fragmentation, collagen accumulation) of the arterial wall. The primary outcomes of structural arterial stiffness will be assessed at baseline and after 3, 6 and 12 months of guideline-based antihypertensive therapy.

SECONDARY OUTCOMES:
Total arterial stiffness measured with pulse wave velocity (m/s) | 12 months
  Local total arterial stiffness measured by tonometry and regional arterial stiffness measured by tonometry. This will be measured at baseline and after 3, 6 and 12 months of guideline-based antihypertensive therapy.
Brachial blood pressure | 12 months
  Upper arm brachial blood blood pressure measurements (mmHg).

OTHER OUTCOMES:
Safety outcome - Acute Kidney Injury | 12 months
  Rise in serum creatinine by at least 50% to a value of >1.5 mg/dL since the last study lab
Safety outcome - Electrolyte abnormalities | 12 months
  Serum sodium <133 or >150 mEq/L, serum potassium <3.0 or >5.5 mEq/L
Safety outcome - Hypotension | 12 months
  Low blood pressure (<90 mmHg systolic) resulting symptoms AND an ER visit or hospitalization.
Safety outcome - Falls | 12 months
  Any fall resulting in an ER visit or hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Gepner, Principal Investigator — William S. Middleton Memorial Veterans Hospital, Madison, WI
Locations (3):
- United States (3):
  - Birmingham VA Medical Center, Birmingham, AL, Birmingham, Alabama
  - Tennessee Valley Healthcare System Nashville Campus, Nashville, TN, Nashville, Tennessee
  - William S. Middleton Memorial Veterans Hospital, Madison, WI, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No